CLINICAL TRIAL: NCT04711408
Title: Virtual Reality During Ultrasound Examination of Women With Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0602-20-TLV
Record Dates: First submitted 2021-01-03; First posted 2021-01-15 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Chronic Pain; Pelvic Pain; Endometriosis
MeSH Terms: conditions — Chronic Pain; Pelvic Pain; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): women allocated to undergo ultrasound for the diagnosis of endometriosis with Virtual reality System
  Interventions: Device: SootheVR: AppliedVR, Los Angeles, California a head-mounted displa
- Standart care (No Intervention): women allocated to undergo ultrasound for the diagnosis of endometriosis without VR

INTERVENTIONS:
Device: SootheVR: AppliedVR, Los Angeles, California a head-mounted displa — For the study group, virtual reality content will be administered to the participant for the duration of the examination through a head-mounted display, RelieVRTM. The VR content for the trial will be "swimming with dolphins".
  Arms: Virtual reality

SUMMARY:
To evaluate the effectiveness of VR as a distraction technique in the management of acute pain and anxiety during ultrasound exam in patients with endometriosis in the outpatient setting.

DETAILED DESCRIPTION:
A prospective, open-label, randomized control trial in a tertiary university-affiliated medical center between April to August 2020. Overall, 100 women will be randomly allocated to undergo ultrasound exam either with the use of VR (study group) or with standard treatment (control group). The primary outcome measures includ self-reported pain, anxiety scores, and vital parameters as pulse rate (PR) and respiratory rate (RR). Pain and anxiety outcomes were measured as numeric rating scores.

ELIGIBILITY:
Inclusion Criteria:

* patient needed ultrasound with the diagnosis of endometriosis. the diagnosis of endometriosis is based on ultrasound finding or previous surgery.

Exclusion Criteria:

* women who reported the use of analgesia 6 hours prior to the procedure

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-06-14 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessments of pain through pain score parameter | 20 minutes
  Assessments of pain through pain score parameter of the NRS questionnaire. Pain will be measured using the Numeric Rating Scale (NRS) which is a 11 point scale from 0 to 10 which is a validated score of measuring pain and anxiety in which 0 is no pain and 10 is the worst imaginable pain and or anxiety.
Assessments of pain through physiological parameters | 10 minutes
  Assessments of pain through physiological parameters of pulse rate. Heart Rate will be measured using Heart Rate-beats per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Lis Maternity Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No